CLINICAL TRIAL: NCT03502148
Title: Phase 1/2, Open-Label, Single-Arm Safety and Efficacy Dose-Finding, Systemic Exposure, and Device Technical Effects of PRV111 (Cisplatin Transmucosal System) in Subjects With Oral Squamous Cell Carcinoma
Brief Title: Safety and Efficacy Study of PRV111 in Subjects With Oral Squamous Cell Carcinoma
Acronym: PRV111
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Privo Technologies (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-001; FD-R-006325 (Other Grant/Funding Number: FDA OOPD); 5R44CA192875-05 (NIH)
Record Dates: First submitted 2018-03-04; First posted 2018-04-18 (Actual); Results first posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-09

CONDITIONS: Oral Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin

STUDY DESIGN:
Intervention Model Description: Phase 1/2, Open-Label, Single-Arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label, Single Arm Study of PRV111 (Experimental): Subjects received 3 treatment applications of PRV111 (Cisplatin Transmucosal System) at each of the 4 planned visits within 3 weeks prior to their tumor surgery.
  Interventions: Drug: PRV111 (Cisplatin Transmucosal System)

INTERVENTIONS:
Drug: PRV111 (Cisplatin Transmucosal System) — Each treatment visit will include one application of a permeation enhancer and then 2, 3 or 5 PRV111 (Cisplatin Transmucosal System) applications depending on the Stage subject is enrolled in.
  Other Names: cisplatin

SUMMARY:
Up to 31 subjects diagnosed with oral squamous cell carcinoma received one application of a permeation enhancer 3 treatment applications of a Cisplatin drug-loaded patch to the tumor site at each of the 4 treatment visits. These 4 treatment visits were scheduled to occur during the 3 weeks prior to the standard of care tumor resection.

Funding Source: FDA OOPD

DETAILED DESCRIPTION:
Up to 31 subjects diagnosed with oral squamous cell carcinoma received one application of a permeation enhancer and 3 treatment applications of a Cisplatin drug-loaded patch to the tumor site at each of 4 treatment visits. These 4 treatment visits were scheduled to occur during the 3 weeks prior to the standard of care tumor resection. After the surgery, subjects were followed for 6 months for disease recurrence.

Ten subjects were enrolled in the study. Up to 21 additional subjects could have been enrolled in Stage 2, if safety and efficacy endpoints were not met. The dose was not changed. All subjects were followed for 6 months post-surgery for disease recurrence.

During and at the conclusion of the treatment period, subjects were monitored for local and systemic safety, tumor response due to the treatment, and systemic drug exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed T1 (<2 cm) or T2 (>2 cm but < or = 4 cm) squamous cell carcinoma (SCC) of the lip or oral cavity (anterior 2/3 of the tongue, floor of mouth, lower and upper gingiva, salivary gland, hard palate, and buccal mucosa).
2. Tumor must be easily accessible, with no evidence of infection or active bleeding, encroaching major vessels or clinical evidence of neural invasion. Not previously irradiated.
3. Tumors must be amenable to surgical resection no later than 21 days post Visit 1.
4. Clinically or radiologically measurable tumor.
5. ECOG Performance Status of < or =2.
6. Adequate renal function as demonstrated by renal creatinine clearance.
7. Adequate organ function as assessed by safety labs.
8. Agree to use effective contraception for 30 days after the last dose of study drug.
9. Absence of any serious medical conditions that would impair the subject's ability to participate.
10. Willing and able to provide written informed consent.
11. Able to return to the study site for treatment and follow-up visits as defined in the protocol.

Exclusion Criteria:

1. Known distal metastasis of the SCC of the oral cavity.
2. Systemic chemotherapy for the treatment of SCC of the head and neck less than 2 years prior to screening.
3. Concurrent documented malignancy, with the exception of localized SCC of the skin.
4. Exposure to any investigational agent within 3 months prior to screening.
5. Known allergy or hypersensitivity to platinum-containing agents.
6. Active, uncontrolled infection requiring systemic therapy.
7. Known or suspected pregnancy, planned pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-10-27 (Actual); Study Completion 2020-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manijeh Goldberg, PhD, Study Director — CEO, Privo Technologies
Locations (5):
- United States (5):
  - Advanced ENT and Allergy, Louisville, Kentucky
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Ben Taub Hospital, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - The University of Texas Health Science Center School of Dentistry, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldberg M, Manzi A, Birdi A, Laporte B, Conway P, Cantin S, Mishra V, Singh A, Pearson AT, Goldberg ER, Goldberger S, Flaum B, Hasina R, London NR, Gallia GL, Bettegowda C, Young S, Sandulache V, Melville J, Shum J, O'Neill SE, Aydin E, Zhavoronkov A, Vidal A, Soto A, Alonso MJ, Rosenberg AJ, Lingen MW, D'Cruz A, Agrawal N, Izumchenko E. A nanoengineered topical transmucosal cisplatin delivery system induces anti-tumor response in animal models and patients with oral cancer. Nat Commun. 2022 Aug 17;13(1):4829. doi: 10.1038/s41467-022-31859-3. PMID 35977936

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-Label, Single Arm Study of PRV111
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects included in the baseline analysis were included in the safety population. Eight subjects were evaluable for the efficacy population.
Groups:
- Open-Label, Single Arm Study of PRV111: Subjects received 3 treatment applications of PRV111 (Cisplatin Transmucosal System) at each of the 4 planned visits (within 3 weeks prior to their tumor surgery). Each treatment included one application of permeation enhancer prior to PRV111 administration.
Arm/Group | Open-Label, Single Arm Study of PRV111
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Age, Continuous [Median (Standard Deviation); unit: years] | 64.3 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Determine an Efficacious Dose (mg/cm2) of PRV111 (Cisplatin Transmucosal System) Via Number of Tumor Responses
Description: The starting dose was 1.5 mg/cm2 of cisplatin. Based on the incidence of dose-limiting toxicities and tumor response, subjects would either continue to receive the starting dose or the dose would be de-escalated to 1.0 mg/cm2 or escalated to 2.5 mg/cm2.
  This measures presents the number of tumor responses during the PRV111 treatment period
Time Frame: Subjects were evaluated for efficacy during the 4 treatment visits in the 21 days prior to surgery
Population: The efficacy population consists of all subjects who completed at least 3 PRV111 treatment visits and met all inclusion/exclusion criteria. The outcome measure is expressed as the count of participants who displayed a tumor response (At least 30% tumor volume reduction based on clinical measurements).
Measure: Count of Participants; unit: Participants
Groups:
- Neoadjuvant PRV111 (Efficacy Population): Subjects who completed at least 3/4 planned PRV111 treatment visits.
Arm/Group | Neoadjuvant PRV111 (Efficacy Population)
Number analyzed (Participants) | 8
Participants | 7

2. Primary Outcome: Determine a Safe Dose (mg/cm2) of PRV111 (Cisplatin Transmucosal System) Via Number of Dose-Limiting Toxicities
Description: The starting dose was 1.5 mg/cm2 of cisplatin. Based on the incidence of dose-limiting toxicities and tumor response, subjects would either continue to receive the starting dose or the dose would be de-escalated to 1.0 mg/cm2 or escalated to 2.5 mg/cm2.
  This measures presents the number of reported dose-limiting toxicities during the PRV111 treatment period
Time Frame: 4 treatment visits in the 21 days prior to surgery
Population: Patients treated with at least 1 PRV111 were included
Measure: Number; unit: dose-limiting toxicities
Groups:
- Neoadjuvant PRV111 (Safety Population): Subjects who received at least a single treatment application of PRV111.
Arm/Group | Neoadjuvant PRV111 (Safety Population)
Number analyzed (Participants) | 10
dose-limiting toxicities | 0

3. Secondary Outcome: Tumor Response (Tumor Volume Change From Baseline and Pre-op Visit, Approximately 21 Days Prior to Surgical Excision of the Tumor)
Description: Assessed by clinical measurement at baseline and at the pre-op visit
Time Frame: Assessed within the 21 days prior to surgical excision of the tumor
Population: Subjects who received at least 3 PRV111 treatments and met all inclusion/exclusion criteria.
Measure: Mean (Full Range); unit: percentage of tumor volume reduction
Arm/Group | Neoadjuvant PRV111 (Efficacy Population)
Number analyzed (Participants) | 8
percentage of tumor volume reduction | 69 [35 to 100]

4. Secondary Outcome: Number of Loco-regional Recurrences
Description: Number of loco-regional recurrences at follow-up
Time Frame: Assessed 1, 3 and 6 months post surgery
Population: Subjects received at least 3 treatment applications of PRV111 (Cisplatin Transmucosal System) at each of the 4 planned visits within 3 weeks prior to their tumor surgery.
Measure: Number; unit: number of locoregional recurrences
Arm/Group | Neoadjuvant PRV111 (Efficacy Population)
Number analyzed (Participants) | 8
number of locoregional recurrences | 0

5. Secondary Outcome: Tumor and Lymph Node (if Available) Platinum Levels
Description: Levels of platinum content in tumor tissue and/or lymph tissue, using a validated bioanalytical ICP-MS method. Resected tissues were digested via microwave and used to evaluate the amount of cisplatin delivered by PRV111 (Correlated to the amount of platinum detected).
Time Frame: 21 days from baseline through surgical excision of the tumor
Measure: Mean (Full Range); unit: µg/g
Arm/Group | Neoadjuvant PRV111 (Safety Population)
Number analyzed (Participants) | 10
µg/g
  Average Tumor Platinum Level | 337 [33 to 1395]
  Average Lymph Node Platinum Level | 110 [11 to 305]

6. Secondary Outcome: Technical Success - Residual Cisplatin Levels Post-application
Description: Platinum content in each residual PRV111, using a validated bioanalytical ICP-MS method and the results for all applications were averaged.
Time Frame: 4 treatment visits in the 21 days prior to surgery
Population: Each patch was analyzed
Measure: Mean (Standard Deviation); unit: percentage of drug released
Arm/Group | Neoadjuvant PRV111 (Safety Population)
Number analyzed (Participants) | 10
percentage of drug released | 91.7 (3.2)

7. Secondary Outcome: Systemic Platinum Levels (Cmax)
Description: Levels of platinum content in blood, using a validated bioanalytical ICP-MS method. Blood drawn was digested via microwave and used to evaluate the amount of systemic cisplatin exposure from PRV111 (Correlated to the amount of platinum detected). A single value for Cmax was calculated by averaging values for all subjects.
Time Frame: Cmax is a single value of the highest concentration of platinum in the blood reported from samples taken post-dose across all 4 treatment visits (Baseline [0], 30, 60, and 120 minutes at Visits 1-4)
Measure: Mean (Full Range); unit: µM
Arm/Group | Neoadjuvant PRV111 (Safety Population)
Number analyzed (Participants) | 10
µM | 0.24 [0.09 to 0.62]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the PRV111 treatment period up to the last follow up visit (up to 6 months post surgery).
Groups:
- Neoadjuvant PRV111 (Safety Population): Subjects received at least 3 treatment applications of PRV111 (Cisplatin Transmucosal System) at each of the 4 planned visits within 3 weeks prior to their tumor surgery.
Arm/Group | Neoadjuvant PRV111 (Safety Population)
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant PRV111 (Safety Population) (N=10)
Failure to Thrive (Metabolism and nutrition disorders) | 1 (1) — This event was reported as severe and not related to study treatment by the investigator. SAE of failure to thrive, which occurred 116 days post last dose of PRV111. The SAE was 124 days after the last administration of PRV111.
Post-Surgical Infected Seroma (Infections and infestations) | 1 (1) — This event was expected from standard of care surgery and determined as possibly related to treatment. The infected seroma followed 2 surgeries, (tumor resection/neck dissection and reconstructive surgery). It resolved with sequelae in the follow-up.
Surgical Complication (Injury, poisoning and procedural complications) | 1 (1) — This event was considered not related to study treatment by the investigator and the event resolved during the follow-up period. The SAE of a procedural complication related to surgery was reported post-operatively 11 days after the last PRV111 dose
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant PRV111 (Safety Population) (N=10)
[During PRV111 Treatment Period] Oral Pain (Gastrointestinal disorders) | 4
[During PRV111 Treatment Period] Glossodynia (Gastrointestinal disorders) | 3
[During PRV111 Treatment Period] Lip Blister (Gastrointestinal disorders) | 2
[During PRV111 Treatment Period] Stomatitis (Gastrointestinal disorders) | 2
[During PRV111 Treatment Period] Constipation (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 2
[During PRV111 Treatment Period] Oral Mucosal Blistering (Gastrointestinal disorders) | 2
[During PRV111 Treatment Period] Tongue Blistering (Gastrointestinal disorders) | 2
[During PRV111 Treatment Period] Tongue Discomfort (Gastrointestinal disorders) | 2
[During PRV111 Treatment Period] Nausea (Gastrointestinal disorders) | 1
[During PRV111 Treatment Period] Angina Pectoris (Cardiac disorders) | 1
[During PRV111 Treatment Period] oropharyngeal pain (Gastrointestinal disorders) | 1
[During PRV111 Treatment Period] salivary duct inflammation (Gastrointestinal disorders) | 1
[During PRV111 Treatment Period] Dysphagia (Gastrointestinal disorders) | 1
[During PRV111 Treatment Period] Swollen Tongue (Gastrointestinal disorders) | 1
[During PRV111 Treatment Period] Gastro Esophageal Reflux Disease (Gastrointestinal disorders) | 1
[During PRV111 Treatment Period] Dry Mouth (Gastrointestinal disorders) | 1
[During PRV111 Treatment Period] Tongue Ulceration (Gastrointestinal disorders) | 1
[During PRV111 Treatment Period] Toothache (Gastrointestinal disorders) | 1
[During PRV111 Treatment Period] Non-cardiac Chest pain (General disorders) | 1
[During PRV111 Treatment Period] Oedema Peripheral (General disorders) | 1
[During PRV111 Treatment Period] Palate Injury (Injury, poisoning and procedural complications) | 1
[During PRV111 Treatment Period] Decreased Appetite (Metabolism and nutrition disorders) | 1
[During PRV111 Treatment Period] Headache (Nervous system disorders) | 1
[During PRV111 Treatment Period] Cough (Respiratory, thoracic and mediastinal disorders) | 1
[Post-PRV111 Treatment, Post-Surgery] Procedural Pain (Injury, poisoning and procedural complications) | 6 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] Procedural Complication (Injury, poisoning and procedural complications) | 3 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] Anxiety (Psychiatric disorders) | 2 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] Constipation (Gastrointestinal disorders) | 2 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] Dysphagia (Gastrointestinal disorders) | 2 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] Malnutrition (Gastrointestinal disorders) | 2 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] Post-Procedural Complication (Injury, poisoning and procedural complications) | 2 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] Nausea (Gastrointestinal disorders) | 2 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] Post Procedural Oedema (Injury, poisoning and procedural complications) | 2 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] Procedural Nausea (Injury, poisoning and procedural complications) | 2 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] Pyrexia (General disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] Infected seroma (Infections and infestations) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] Fatigue (General disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] post operative hypertension (Injury, poisoning and procedural complications) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] skin graft failure (Injury, poisoning and procedural complications) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] weight decreased (Investigations) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] fluid overload (Metabolism and nutrition disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] hyperglycemia (Metabolism and nutrition disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] hypervolemia (Metabolism and nutrition disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] hypophosphatemia (Metabolism and nutrition disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] lactic acidosis (Metabolism and nutrition disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] malnutrition (Metabolism and nutrition disorders) | 2 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] dysarthria (Nervous system disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] agitation (Psychiatric disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] insomnia (Psychiatric disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] urinary retention (Renal and urinary disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] productive cough (Respiratory, thoracic and mediastinal disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] skin disorder (Skin and subcutaneous tissue disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] swelling face (Skin and subcutaneous tissue disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] hypotension (Vascular disorders) | 1 — post-PRV111 treatment period; post-surgery
[Post-PRV111 Treatment, Post-Surgery] shock (Vascular disorders) | 1 — post-PRV111 treatment period; post-surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT03502148/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT03502148/SAP_001.pdf
  • Informed Consent Form (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT03502148/ICF_002.pdf